CLINICAL TRIAL: NCT00798486
Title: In-Clinic Evaluation of the Redwood A1c Test Kit With Lay-Users and Professionals
Brief Title: Evaluation of the A1CNow+ Test Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2008-14
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with and without Diabetes (Other): Subjects participating in this study included 93 who had diabetes and 17 who did not have diabetes.
  Interventions: Device: A1C Test Kit

INTERVENTIONS:
Device: A1C Test Kit — Subjects tested 3 times with A1C test kits. Two tests were performed by the subject and the third test was performed by a healthcare professional (HCP). All results were compared to results from a laboratory glucose analyzer (TOSOH).
  Other Names: A1CNow SELFCHECK

SUMMARY:
The purpose of this study was to assure that consumers can successfully use the new version of A1CNow+ along with revised instructional materials.

DETAILED DESCRIPTION:
The purpose of this study was to assure that consumers could successfully use the new version of A1CNow+ Test Kit along with revised instructional materials. The primary objective was to establish accuracy and secondary objectives were to establish precision, comprehension of instructional materials, and user feedback about the overall testing experience.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18 and older) approximately 80% being ≤55 years old
2. Persons with:

   * known diabetes (type 1 or type 2) and pre-diabetes - approximately 85% of subject population per site
   * no known diagnosis of diabetes - approximately 15% of subject population per site
3. Individuals who are interested in performing a test using the kit at home
4. Individuals willing to complete all study procedures (including venous draw and allowing site staff to perform finger punctures)
5. Individuals who are able to speak, read, and understand English
6. Individuals able to read out loud the first 5 lines of the A1C Test Kit instructional materials to demonstrate ability to read the print (may use glasses, if needed)

Exclusion Criteria:

1. Individuals taking prescription anticoagulants (such as Warfarin or heparin) or have clotting problems that may prolong bleeding. (Taking Plavix or aspirin daily is not excluded)
2. Individuals with known Rheumatoid Arthritis or other condition causing significant impairment of manual dexterity
3. Individuals with a known hemoglobin variant such as HbS or HbC
4. Individuals with any known disorder of the blood or blood-forming organs (such as recovery from blood loss, hemolytic anemia, or iron deficiency anemia)
5. Individuals who have received a blood transfusion within the 4 months prior to the study.
6. Persons with known infection with a bloodborne pathogen (e.g. HIV, hepatitis)
7. Individuals working for a competitive medical device company
8. Individuals who have participated in previous studies on the A1CNow+ product
9. Persons missing a digit or partial digits on the hand
10. Individuals with the following impairments which, in the opinion of the investigator, would seriously compromise the integrity of the study:

    * Significant visual impairment
    * Significant hearing impairment
    * Cognitive disorder
    * Any other condition as per investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chang, MD, Principal Investigator — John Muir Physician Network Clinical Research Center; Joy Frank, RN, Principal Investigator — Consumer Products Testing
Locations (2):
- United States (2):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Consumer Product Testing Co., Inc., Fairfield, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With and Without Diabetes
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 110
Age, Continuous [Median (Full Range); unit: years] | 46 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 70
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of A1C Results Either Equal To Or Within +/- 13.5% of the Laboratory Method (ACCURACY)
Description: This outcome measure reports the number of A1c test results for which the percent difference (absolute value) between results from the subject meter and the laboratory method was less than or equal to 13.5%.
Time Frame: One hour
Measure: Number; unit: number of A1c results
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 110
number of A1c results
  Subjects had DVD and Written Instructions (n=101) | 94
  Subjects had Written Instructions only (n=77) | 71

2. Secondary Outcome: Average Within Subject Coefficient of Variation CV (PRECISION)
Description: The average Coefficient of Variation (CV) was computed by calculating the square of the CV for each pair of A1c self-test results, averaging this square value over the number of subjects included in the analysis, and then taking the square root.
Time Frame: One hour
Population: Precision Coefficient of Variation (CV)was analyzed using meter results from subject data that had numeric values for duplicate A1c self-tests. Subject data was not used in this outcome measure analysis when there had been a protocol deviation or when one (or both) A1c self-tests resulted in an error code.
Measure: Number; unit: average percentage CV
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 74
average percentage CV | 4.57

3. Secondary Outcome: Percentage of Subjects Who Experienced First Time Failures (FTF) During Testing
Description: For the comprehension analysis, subjects were divided into 2 groups. One group (n=56 subjects) was given both written (Quick Reference Guide) and DVD instruction material. The other group (n=54 subjects) was given only written instruction material. First time failure (FTF) was defined as:
  * The subject could not use the product without HCP assistance.
  * The subject could not complete the test. User error rendered one or more parts unusable.
  * The subject completed the test after one or more mistakes; the result was an error code instead of a numerical value.
Time Frame: One hour
Measure: Number; unit: percentage of subjects
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 110
percentage of subjects
  Subjects had DVD and Written Instructions | 11
  Subjects had Written Instructions Only | 40

4. Secondary Outcome: Number of Participants Who Provided These Ratings For Overall Testing Experience With A1C Test Kit
Description: Subjects rated features of the A1C Test Kit, including 'Overall Testing Experience'. The rating scale was 4 (Excellent) to 1 (Poor).
Time Frame: One hour
Measure: Number; unit: number of participants
Arm/Group | Subjects With and Without Diabetes
Number analyzed (Participants) | 110
number of participants
  4 - Excellent | 65
  3 - Very Good | 38
  2 - Good | 7
  1 - Poor | 0

ADVERSE EVENTS:
Arm/Group | Subjects With and Without Diabetes
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less